CLINICAL TRIAL: NCT03444337
Title: High-resolution Contrast-Enhanced MRI of Atrial Fibrillation Patients Prior to FIRM Ablation
Brief Title: High-resolution MRI of Atrial Fibrillation Patients Prior to Focal Impulse and Rotor Modulation (FIRM) Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, John Hummel, Professor of Internal Medicine, Ohio State University
Other Study IDs: 2016H0200
Record Dates: First submitted 2018-02-18; First posted 2018-02-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: ablation; atrial fibrillation; FIRM
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Catheter Ablation Group: Patients undergoing FIRM guided ablation of paroxysmal or persistent atrial fibrillation with pre-procedure high resolution cardiac MRI
  Interventions: Device: Catheter Ablation

INTERVENTIONS:
Device: Catheter Ablation

SUMMARY:
Patients undergoing FIRM guided ablation of atrial fibrillation will undergo high resolution MRI imaging to determine correlation of underlying anatomic fibrotic regions with FIRM targeted sites for ablation.

DETAILED DESCRIPTION:
The project will be a prospective trial involving patients consented for a clinically indicated atrial fibrillation (AF) ablation using FIRM mapping. The purpose of the study is to collect additional information before, during, and after the ablation procedure. All patients will undergo a contrast-enhance MRI scanning with gadolinium-based contrast agent prior to the procedure as it provides a 3-dimensional image of both the left atria and right atria. The primary endpoint of this study will be the presence or absence of a correlation between micro-anatomic fibrotic tracks, determined by a combination of atrial wall thickness, and local scar and fibrosis, and sites of FIRM map indicated rotor activity. Medical information will also be collected after the patients 2nd, 3rd and 6 month standard of care doctor visits. There are no additional risks associated with this protocol over and above that of the standard risk of atrial fibrillation ablation with FIRM, and those associated with the standard risk of magnetic resonance imaging with gadolinium contrast agent, but there is a small risk of the loss of confidentiality when participating in an observational study. The potential benefits includes the possibility of greater understanding of the patient's specific disease state.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic paroxysmal or persistent atrial fibrillation undergoing clinically-indicated ablation procedure employing FIRM mapping with pre-operative MRI.
2. Subjects must be at least 18 years of age.

Exclusion Criteria:

1. LAA thrombus present on pre-procedure TEE
2. Unable to undergo MRI imaging
3. Unable to receive gadolinium contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic paroxysmal or persistent atrial fibrillation undergoing clinically-indicated ablation procedure employing FIRM mapping with pre-operative MRI
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-11-03 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of FIRM targeted sites with MRI fibrotic regions | Immediate post-procedure analysis
  The primary endpoint of this study will be the presence or absence of a correlation between micro-anatomic fibrotic tracks of reentry, determined by a combination of atrial wall thickness, and local scar and fibrosis, and sites of FIRM map indicated rotor activity.

SECONDARY OUTCOMES:
Success or failure of electrical isolation of PV | Immediate post-procedure
  PV analysis by intra-cardiac recordings to determine PV isolation
Termination of AF or significant slowing of AF | Immediate post-procedure
  Incidence of early termination or >10% increase in AF cycle length at the site of FIRM detected rotor formation and whether there is a correlation with fibrotic scar.
Correlation of recurrence of AF six months post ablation with percentage of fibrosis ablated | Six months post ablation
  Correlation of recurrence of AF six months post ablation with percentage of fibrosis ablated
e. Correlation of absence atrial tachycardia or atrial flutter 6 months post ablation with connection of FIRM sites to areas of fibrotic scar or anatomic barriers. | Six months post-ablation
  e. Correlation of absence atrial tachycardia or atrial flutter 6 months post ablation with connection of FIRM sites to areas of fibrotic scar or anatomic barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Golden-Kreutz, RN, Phd, Study Director — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No